CLINICAL TRIAL: NCT05911776
Title: Nasal Packing Versus Intravenous Dexmedetomidine in Turbinate Surgeries: A Randomized Double-Blinded Trial
Brief Title: Nasal Packing Versus Intravenous Dexmedetomidine in Turbinate Surgeries
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Gamal Hendawy Shams, Lecturer of Anesthesiology, Surgical Intensive Care and Pain Medicine Faculty of Medicine Kafr-El Sheikh University, Kafrelsheikh University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KFSIRB200-3
Record Dates: First submitted 2023-05-18; First posted 2023-06-22 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Nasal Packing; Dexmedetomidine; Turbinate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group NP (nasal packing Dexmedetomidine) (Active Comparator): Patients will receive nasal packing Dexmedetomidine (1.5 μg/kg intranasal dexmedetomidine diluted with saline) and Intravenous infusion saline.
  Interventions: Drug: Nasal packing Dexmedetomidine
- Group IV (Intravenous Dexmedetomidine) (Active Comparator): Patients will receive 0.5 μg/kg bolus over 10 min then 0.1- 0.4 μg/kg IV infusion Dexmedetomidine and nasal packing with saline.
  Interventions: Drug: Intravenous Dexmedetomidine

INTERVENTIONS:
Drug: Nasal packing Dexmedetomidine — patients will receive nasal packing Dexmedetomidine (1.5 μg/kg intranasal dexmedetomidine diluted with saline) and Intravenous infusion saline.
  Arms: Group NP (nasal packing Dexmedetomidine)
Drug: Intravenous Dexmedetomidine — patients will receive 0.5 μg/kg bolus over 10 min then 0.1- 0.4 μg/kg Intravenous infusion Dexmedetomidine and nasal packing with saline.
  Arms: Group IV (Intravenous Dexmedetomidine)

SUMMARY:
Comparing of nasal packing DEX and IV DEX for controlling the intraoperative bleeding after turbinate surgery.

DETAILED DESCRIPTION:
Dexmedetomidine (DEX) is a highly selective α2 adreno-receptor agonist with higher affinity to a2 adreno-receptor than clonidine, and this makes DEX primarily sedative and anxiolytic. The elimination half-life of DEX (t1/2b) is 2 h and the redistribution half-life (t1/2a) is 6 min, and this short half-life makes it an ideal drug for intravenous titration. Potentially desirable effects include decreased requirements for other anesthetics and analgesics.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 65 years
* Both sexes
* American Society of Anesthesiologists (ASA) physical status classification I or II.
* Undergo turbinate surgery

Exclusion Criteria:

* Patients with a body mass index > 30 kg/m2 existing or recent significant disease.
* Contraindications to the use of dexmedetomidine .
* History or presence of a significant disease significant cardiovascular disease risk factors.
* Significant coronary artery disease or any known genetic predisposition.
* History of any kind of drug allergy,
* Drug abuse.
* Clinically significant abnormal findings in physical examination, electrocardiographic (ECG) or laboratory screening.
* Known systemic disease requiring the use of anticoagulants,
* Patients with a history of previous turbinate surgery.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-06-30 (Actual); Primary Completion 2024-02-27 (Actual); Study Completion 2024-02-27 (Actual)

PRIMARY OUTCOMES:
Amount of intraoperative blood loss | Intraoperative up to 6hours
  Measuring the volume of suctioned blood in graduated columns, which will contain an anticoagulant to prevent coagulation and clotting and weighing gauze sponges.

SECONDARY OUTCOMES:
Pain score | 24 hours postoperative
  Visual analogue scale (VAS) (0, no discomfort and no pain; 10, a high level of discomfort and maximum pain)
Quality of intraoperative surgical field | Intraoperative up to 6hours
  Quality of intraoperative surgical field during after turbinate surgery will be evaluated by the surgeons by rating the amount of bleeding according to a 6-point scale by Formmer's scores of surgical field quality (0= no bleeding; 1= bleeding, so mild it was not even a surgical nuisance; 2= moderate bleeding, a nuisance but without interference; 3= moderate bleeding that moderately compromised surgical; 4= bleeding, heavy but controllable, that significantly interfered; 5= massive uncontrollable bleeding)
Patient's general satisfaction | 24 hours postoperative
  Patients' satisfaction will be measured immediately postoperative and using a five-point Likert scale consisting of "very dissatisfied," "dissatisfied," "unsure," "satisfied," and "very satisfied.

CONTACTS AND LOCATIONS:
Locations (1):
- Karelsheikh University Hospital, Kafr ash Shaykh, Karelsheikh, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon reasonable request from the corresponding author for one year after study completion.
Supporting Information: Study Protocol